CLINICAL TRIAL: NCT04444778
Title: Intermitent Hypoxia and Its Pathophysiology Consequences in the Sleep Apnea-Hypopnea Syndrome. Basic, Clinical and Therapeutically Study.
Brief Title: Intermitent Hypoxia and Its Pathophysiology Consequences in the Sleep Apnea-Hypopnea Syndrome.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Alberto Alonso Fernandez (Other Government)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Alberto Alonso Fernandez, Principal investigator, Fundació d'investigació Sanitària de les Illes Balears
Organization: Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI19/00875
Record Dates: First submitted 2020-06-06; First posted 2020-06-24 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Sleep Apnea, Obstructive
Keywords: sleep apnea syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous positive airway pressure (Active Comparator): Diet and general life style recommendations plus continuous positive airway pressure (CPAP).
  Interventions: Device: CPAP
- Conservative treatment (No Intervention): Diet and general life style recommendations.

INTERVENTIONS:
Device: CPAP — Continuous positive airway pressure
  Arms: Continuous positive airway pressure

SUMMARY:
Clinical trial on the effect of continuous positive pressure (CPAP). Objectives: 1) To assess the total or partial recovery of oxidative and inflammatory damage after recovering IH. 2) To check whether the results obtained in vitro on the recovery of the damage according to the form of manifestation of IH are validated in SAHS patients. 3) To determine if CPAP reduces nighttime blood pressure and arterial stiffness depending on whether or not patients have a non-dipping pattern of blood pressure and depending on the degree of correction of IH. 4) To clarify whether residual nocturnal hypoxemia influences the recovery of oxidative and inflammatory damage in patients. 5) To determine nasal and intestinal microbioma and the effect of CPAP treatment

DETAILED DESCRIPTION:
Design: Randomized, parallel group, non-blinded, controlled clinical trial compared with conventional treatment.

A. Protocol and intervention Patients with an AHI>30 h-1 will be assigned, using a 1:1 randomization table, to lifestyle recommendations treatment or to lifestyle recommendations plus nasal CPAP, for a period of 4 months. CPAP pressure will be titled with automatic using an AutoSet II device, ResMed.

B. Sample size For the estimation of the sample size, previous data from our group were used. In this case, in order to compare the effect of CPAP in a subgroup of patients with well-controlled OSA and in another with residual hypoxemia; it would be necessary to randomize a total of 85 patients with OSA.

C. Ethical considerations

* Indication of CPAP treatment for the prevention of cardiovascular morbidity and mortality in OSA patients without daytime sleepiness is not yet accepted.
* Those patients with a urgent study indication for the diagnosis and treatment of respiratory sleep disorders (professional drivers, respiratory failure or risk professions) will be excluded from the project. In the other cases, the delay in healthcare for the performance of Polysomnography and CPAP titration exceeds the duration of the study, therefore that patients assigned to the control arm (conventional treatment) will not be exposed to a higher risk than the general population.

D. Methods

* Polysomnography. It will be used as a screening test previous the randomization of the included patients. The exploration and its interpretation will be carried out following the recommendations of the American Academy of Sleep Medicine. Based on the results of this test, only those patients with an AHI will continue in the study when AHI >30 h-1. In these patients the determinations listed below will be carried out immediately before randomization (visit 1), at 4 weeks (visit 2), 16 weeks (visit 4) of allocation to the corresponding treatment group
* Clinical data: The medication used and other associated diseases already diagnosed will be recorded.
* Vital signs: recording of blood pressure, by means of a conventional triple taking, and heart rate.
* Anthropometric characteristics: age and weight in basal conditions, the perimeter of the neck and waist / hip index will be measured. The lean mass index will be determined using a Bodystat 1500 impedance system (Bodystat Ltd, United Kingdom).
* Questionnaires: Epworth Sleepiness Scale, generic health-related quality of life (SF-12 and EuroQoL) and daily physical activity (International Physical Activity Questionnaire or iPAQ).
* Laboratory findings: blood count, coagulation, creatinine, serum sodium and potassium; glycated hemoglobin (HbA1c) and blood glucose and insulin levels in fasting, from these values will determine the resistance and sensitivity to insulin using the HOMA and QUICKI indices; total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides; and troponin I, homocysteine, NT-pro BNP and highly sensitive C-reactive protein.
* Blood venous samples. 20 mL of venous blood will be collected, storing the plasma obtained at -80 ºC for subsequent determination of inflammatory markers (IL-1ß, IL-6, IL-8, HIF 1- 'NF * + and TNF-a), oxidative stress (8-isoprostane), endothelial damage (endothelin, angiotensin II, VCAM-1 and ICAM-1), of sympathetic activity (neuropeptide Y, metanephrines) and appetite-regulating hormones (leptin and adiponectin).
* Plasma proteins from peripheral blood samples will be analyzed using a high-throughput multiplex immunoassay technology based on the Proximity Extension Assays (PEA) (OLINK Bioscience, Uppsala, Sweden). Olink (OLINK Bioscience, Uppsala, Sweden).
* Night pulse oximetry. To assess the existence of residual nocturnal hypoxemia.
* Arterial stiffness. According to the recommendations by Sphygmo-Corsystem (version 7, AtCor Medical, Sydney, Australia).
* Study of the gut and pharyngeal microbiota by massive sequencing (next generation sequencing) after PCR amplification of the 16S rRNA gene, paired-end sequencing with Illumina technology (16S Amplicon and XT Nextera Metagenomic) and subsequent metataxonomic analysis of the microbial populations.
* Ambulatory blood pressure monitoring (ABPM) with Mortara's Ambulo 2400 ambulatory blood pressure device.
* In the patients assigned to the CPAP treatment arm, a count of the hours of use of the CPAP will be carried out at each visit by directly reading the automatic counter of each equipment.

Statistic analysis The data will be expressed as mean ± standard deviation, median (interquartile range) or percentage, depending on their type and distribution. For comparison between groups Student's t-test, the U-Mann-Whitney or the chi-square test will be used, as appropriate. The relations between variables will be analyzed using Pearson's correlation and multiple linear regression analysis. The effect of treatment will be evaluated using general linear models and repeated measures analysis of variance, with multiple comparisons post-hoc using the Bonferroni test. A multiple logistic regression model will be applied to determine the related variables with a response to treatment. Values of p <0.05 will be considered statistically significant. The statistical study will be performed with the SPSS program version 15.0.

ELIGIBILITY:
Inclusion Criteria:

* Cases: patients with AHI > 30
* Controls: subjects with AHI < 5 and Epworth >10

Exclusion Criteria:

* Epworth>18
* BMI<40Kg/M2
* Arterial Hypertension
* Mellitus Diabetes
* Cerebrovascular disease
* Ischemic heart disease
* Cardiac arrhythmia
* Chronic cardiovascular diseases
* Daytime Oxygen saturation>95%
* Risk professions (professional drivers)
* Concomitant treatment with antihypertensives, statins, antidiabetics, beta-blockers or systemics corticosteroids.
* Pretreatment with CPAP.
* Participation in another clinical trial thirty days prior to randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-05-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 8 isoprostane levels | 4 months
  To compare the change in 8 isoprostane levels between the patients allocated to CPAP group and the control group
Change from baseline in microbiota population diversity from stool samples | 4 months
  To compare the change in in microbiota population diversity, after massive sequencing and amplification of the 16S rRNA gene from stool samples between the patients allocated to CPAP group and the control group
Change from baseline in microbiota population diversity from nasopharyngeal samples | 4 months
  To compare the change in microbiota population diversity, after massive sequencing and amplification of the 16S rRNA gene from nasopharyngeal samples between the patients allocated to CPAP group and the control group
Change from baseline in microbiota population abundance from stool samples | 4 months
  To compare the change in microbiota population abundance, after massive sequencing and amplification of the 16S rRNA gene from stool samples between the patients allocated to CPAP group and the control group
Change from baseline in microbiota population abundance from nasopharyngeal samples | 4 months
  To compare the change in microbiota population abundance, after massive sequencing and amplification of the 16S rRNA gene from nasopharyngeal samples between the patients allocated to CPAP group and the control group
Change from baseline in microbiota population color maps from stool samples | 4 months
  To compare the change in microbiota population color maps, after massive sequencing and amplification of the 16S rRNA gene from stool samples between the patients allocated to CPAP group and the control group
Change from baseline in microbiota color maps from nasopharyngeal samples | 4 months
  To compare the change in microbiota population color maps, after massive sequencing and amplification of the 16S rRNA gene from nasopharyngeal samples between the patients allocated to CPAP group and the control group

SECONDARY OUTCOMES:
Augmentation index (%) | Baseline and 4 months
  To compare Augmentation index (%) in OSA and in non-OSA patients, and the change from baseline between the patients allocated to CPAP group and the control group.
Pulse wave velocity (m/sec) | Baseline and 4 months
  To compare pulse wave velocity (m/sec) in OSA and in non-OSA patients, and the change from baseline between the patients allocated to CPAP group and the control group.
Aortic systolic blood pressure central (mmHg) | Baseline and 4 months
  To compare systolic blood pressure central (mmHg) in OSA and in non-OSA patients, and the change from baseline between the patients allocated to CPAP group and the control group.
Diastolic blood pressure central (mmHg) | Baseline and 4 months
  To compare diastolic blood pressure central (mmHg) in OSA and in non-OSA patients, and the change from baseline between the patients allocated to CPAP group and the control group.
Subendocardial viability ratio (%) | Baseline and 4 months
  To compare subendocardial viability ratio (%) in OSA and in non-OSA patients, and the change from baseline between the patients allocated to CPAP group and the control group.
Central augmentation pressure (mmHg) | Baseline and 4 months
  To compare central augmentation pressure (mmHg) in OSA and in non-OSA patients, and the change from baseline between the patients allocated to CPAP group and the control group.
Time to reflection (ms) | Baseline and 4 months
  To compare time to reflection (ms) in OSA and in non-OSA patients, and the change from baseline between the patients allocated to CPAP group and the control group.
Peripheral systolic blood pressure (mmHg) | Baseline and 4 months
  To compare peripheral systolic blood pressure (mmHg) in OSA and in non-OSA patients, and the change from baseline between the patients allocated to CPAP group and the control group.
Peripheral diastolic blood pressure (mmHg) | Baseline and 4 months
  To compare diastolic blood pressure central (mmHg) in OSA and in non-OSA patients, and the change from baseline between the patients allocated to CPAP group and the control group.
Nocturnal blood pressure dipping | Baseline and 4 months
  To compare number of patients with nocturnal blood pressure dipping in OSA and in non-OSA patients, and the change from baseline between the patients allocated to CPAP group and the control group.
Nocturnal hypertension. | Baseline and 4 months
  To compare number of patients with nocturnal hypertension in OSA and in non-OSA patients, and the change from baseline between the patients allocated to CPAP group and the control group.
Patients with undiagnosed hypertension | Baseline and 4 months
  To compare number of patients with undiagnosed hypertension in OSA and in non-OSA patients, and the change from baseline between the patients allocated to CPAP group and the control group.
C-reactive protein (CRP) | Baseline and 4 months
  To compare CRP in OSA and in non-OSA patients, and the change from baseline between the patients allocated to CPAP group and the control group.
Homocysteine | Baseline and 4 months
  To compare homocysteine (μmol/L) in OSA and in non-OSA patients, and the change from baseline between the patients allocated to CPAP group and the control group.
Endothelin | Baseline and 4 months
  To compare endothelin levels in OSA and in non-OSA patients, and the change from baseline between the patients allocated to CPAP group and the control group.
8 isoprostane levels in OSA and in non-OSA patients | Baseline
  To compare 8 isoprostane levels in OSA and in non-OSA patients.
Lipid profile | Baseline and 4 months
  To compare lipid profile with same units of measure (all in mg/dL) in OSA and in non-OSA patients and to compare baseline (OSA vs. non-OSA), and the change from baseline in lipid profile between the patients allocated to CPAP group and the control group.
Circulating inflammatory proteomic profile in OSA | Baseline and 4 months
  To compare the circulating inflammatory proteomic profile using proximity expression assay technology (Olink®, Sweden, which comprised 96 proteins. All data are expressed as normalized protein expression values) in OSA and in non-OSA patients and to compare the change from baseline the circulating inflammatory proteomic profile between the patients allocated to CPAP group and the control group.
Systemic inflammation. | Baseline and 4 months
  To compare systemic inflammation (IL-6, IL-8, TNF-1alpha) with same units of measure (all in pg/mL) in OSA and in non-OSA patients and to compare the change from baseline between the patients allocated to CPAP group and the control group.
Intake-regulating hormones. | Baseline and 4 months
  To compare intake-regulating hormones with same units of measure (all in µg/mL) in OSA and in non-OSA patients and to compare the change from baseline between the patients allocated to CPAP group and the control group.
Change from baseline in number of patients with desaturation index >3% | 4 months
  To compare the change from baseline in number of patients with desaturation index >3% between the patients allocated to CPAP group and the control group
Microbiota population abundance from stool and nasopharyngeal samples in OSA and in non-OSA patients | Baseline
  To compare microbiota population abundance from stool and nasopharyngeal samples in OSA and in non-OSA patients
Microbiota population diversity from stool and nasopharyngeal samples in OSA and in non-OSA patients | Baseline
  To compare microbiota population diversity from stool and nasopharyngeal samples in OSA and in non-OSA patients
Microbiota population color maps from stool and nasopharyngeal samples in OSA and in non-OSA patients | Baseline
  To compare microbiota population color maps from stool and nasopharyngeal samples in OSA and in non-OSA patients
Relationships of microbiota population diversity from stool and nasopharyngeal samples in OSA to blood pressure profile. | Baseline and 4 months
  To relate microbiota population diversity from stool and nasopharyngeal samples to blood pressure profile.
Relationships of microbiota population abundance from stool and nasopharyngeal samples in OSA to blood pressure profile | Baseline and 4 months
  To relate microbiota population diversity from stool and nasopharyngeal samples to blood pressure profile.
Relationships of microbiota population color maps from stool and nasopharyngeal samples in OSA to blood pressure profile | Baseline and 4 months
  To relate microbiota population color maps from stool and nasopharyngeal samples to blood pressure profile.
Relationships of microbiota population diversity from stool and nasopharyngeal samples in OSA to augmentation index. | Baseline and 4 months
  To relate microbiota population diversity from stool and nasopharyngeal samples to augmentation index.
Relationships of microbiota population abundance from stool and nasopharyngeal samples in OSA to augmentation index. | Baseline and 4 months
  To relate microbiota population diversity from stool and nasopharyngeal samples to augmentation index.
Relationships of microbiota population color maps from stool and nasopharyngeal samples in OSA to augmentation index. | Baseline and 4 months
  To relate microbiota population color maps from stool and nasopharyngeal samples to augmentation index.
Relationships of microbiota population diversity from stool and nasopharyngeal samples in OSA to pulse wave velocity. | Baseline and 4 months
  To relate microbiota population diversity from stool and nasopharyngeal samples to pulse wave velocity.
Relationships of microbiota population abundance from stool and nasopharyngeal samples in OSA to pulse wave velocity. | Baseline and 4 months
  To relate microbiota population diversity from stool and nasopharyngeal samples to pulse wave velocity.
Relationships of microbiota population color maps from stool and nasopharyngeal samples in OSA to pulse wave velocity. | Baseline and 4 months
  To relate microbiota population color maps from stool and nasopharyngeal samples to pulse wave velocity.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Alonso, Dr, Principal Investigator — Fundació d'investigació Sanitària de les Illes Balears
Locations (2):
- Spain (2):
  - Hospital Son Espases, Palma, Balearic Islands
  - Hospital Son Llatzer, Palma, Balearic Islands

IPD SHARING:
Plan to Share IPD: No